CLINICAL TRIAL: NCT07204587
Title: A Stratified, Partially Randomized Study Comparing Autologous Semitendinosus Tendon Graft and Meniscal Allograft Transplantation in Young Adults With Post-Meniscectomy Syndrome
Brief Title: Semitendinosus Autograft vs Meniscal Allograft in Post-Meniscectomy Syndrome
Acronym: MAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChangGungMH MeniscusTransplant
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: Meniscal Injuries; Meniscal Tear; Meniscus Lesion
Keywords: meniscal allograft; autologous tendon graft; Post-meniscectomy syndrome; Meniscus deficiency

STUDY DESIGN:
Intervention Model Description: This study uses a stratified, partially randomized parallel assignment model. Eligible patients are allocated into four groups: randomized autologous semitendinosus tendon graft, randomized meniscal allograft transplantation, patient-preference autologous tendon graft, and patient-preference meniscal allograft transplantation. Even in the randomized groups, participants retain the option to switch to their preferred treatment after allocation, ensuring both methodological rigor and ethical feasibility. This design allows assessment of comparative outcomes under randomized conditions as well as in real-world preference-based clinical practice.
Who Masked: Outcomes Assessor
Masking Description: Postoperative MRI and patient-reported outcome measures (PROMs) will be evaluated by independent assessors blinded to treatment allocation. Participants, surgeons, and investigators will be aware of the intervention due to the surgical nature of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 Autologous Semitendinosus Tendon Graft (Randomized) (Experimental): Patients randomized to this arm will undergo meniscal reconstruction using autologous semitendinosus tendon grafts (diameter ≥ 6 mm). Standard two-tunnel fixation technique will be applied, with Fibertape internal brace augmentation. ACL reconstruction may be performed simultaneously if indicated.
  Interventions: Procedure: Autologous Semitendinosus Tendon Graft
- A2 Meniscal Allograft Transplantation (Randomized) (Experimental): Patients randomized to this arm will receive size-matched fresh-frozen meniscal allografts. Fixation will be performed using the standard two-tunnel technique.
  Interventions: Procedure: Meniscal Allograft Transplantation (MAT)
- Meniscal Allograft Transplantation (Patient Preference) (Experimental): Patients who decline randomization but choose allograft transplantation will undergo the same surgical procedure as Arm A2, with fresh-frozen meniscal allografts.
  Interventions: Procedure: Meniscal Allograft Transplantation (MAT)
- Autologous Semitendinosus Tendon Graft (Patient Preference) (Experimental): Patients who decline randomization but choose autologous tendon grafting will undergo the same procedure as Arm A1, using semitendinosus tendon grafts with Fibertape internal brace augmentation.
  Interventions: Procedure: Autologous Semitendinosus Tendon Graft

INTERVENTIONS:
Procedure: Autologous Semitendinosus Tendon Graft — Meniscal reconstruction will be performed using autologous semitendinosus tendon harvested from the ipsilateral leg. The graft diameter must be at least 6 mm. A two-tunnel fixation technique will be employed, securing the graft to the tibial plateau at the anatomic meniscal root sites. The graft will be shaped and positioned to mimic the native meniscal contour. Fibertape internal brace augmentation will be added to enhance fixation strength and graft stability. If concomitant anterior cruciate ligament reconstruction is indicated, the graft choice and ACL technique will be determined by the surgeon, without restriction. Postoperative rehabilitation will follow a standardized protocol across all centers.
  Arms: A1 Autologous Semitendinosus Tendon Graft (Randomized); Autologous Semitendinosus Tendon Graft (Patient Preference)
Procedure: Meniscal Allograft Transplantation (MAT) — Meniscal allograft transplantation will use size-matched, fresh-frozen allograft menisci prepared according to institutional tissue bank standards. Grafts will be fixed using a two-tunnel bone plug technique, restoring the anatomic root insertions. The allograft will be centrally positioned within the tibiofemoral compartment, and centralization sutures may be added at the discretion of the operating surgeon. All procedures will be standardized across participating centers, and postoperative rehabilitation protocols will be identical to those used in the autologous graft arm.
  Arms: A2 Meniscal Allograft Transplantation (Randomized); Meniscal Allograft Transplantation (Patient Preference)

SUMMARY:
This multicenter, stratified, partially randomized clinical trial aims to compare autologous semitendinosus tendon graft and meniscal allograft transplantation (MAT) in young adults with post-meniscectomy syndrome. The meniscus plays a critical role in load distribution, shock absorption, and joint stability. After meniscectomy, insufficient meniscal tissue often leads to persistent pain, swelling, and functional decline, increasing the risk of early osteoarthritis.

Two reconstructive strategies are clinically available: MAT provides immediate biomechanical function but requires donor matching and carries higher costs, while autologous tendon graft offers stable supply and no immunologic risk but lacks long-term clinical validation.

In this study, 40 patients aged 18-45 years will be enrolled. Participants will be allocated into four groups (randomized MAT, randomized autograft, patient-preference MAT, patient-preference autograft). All procedures will use a two-tunnel fixation technique with additional internal brace support.

The primary endpoint is the improvement in KOOS (Knee Injury and Osteoarthritis Outcome Score) at 24 months postoperatively. Secondary endpoints include MRI-based assessment of graft morphology and extrusion, reoperation rate, complications, patient satisfaction, and return-to-sport time.

This trial will provide critical evidence regarding the comparative effectiveness and feasibility of tendon autograft versus meniscal allograft in real-world clinical settings, potentially informing surgical decision-making and future treatment guidelines for post-meniscectomy syndrome.

DETAILED DESCRIPTION:
Post-meniscectomy syndrome represents a challenging condition in young adults, characterized by persistent pain, swelling, and functional impairment after partial or subtotal meniscectomy. The lack of sufficient meniscal tissue predisposes patients to abnormal tibiofemoral loading and early onset osteoarthritis. Current reconstructive options remain limited, and there is no consensus on the optimal surgical strategy.

Meniscal allograft transplantation (MAT) has been the most widely accepted method, offering immediate restoration of meniscal morphology and load-distributing capacity. However, MAT is constrained by donor availability, graft costs, and local regulations. In contrast, autologous tendon grafts-most commonly using semitendinosus-are readily available, carry no risk of rejection, and reduce cost barriers. Early biomechanical and translational studies suggest that autologous tendon grafts may adapt to meniscal-like properties, yet long-term clinical data remain scarce.

This trial employs a stratified, partially randomized design to balance methodological rigor with patient autonomy and ethical feasibility. Participants are assigned to autologous tendon graft or MAT either through randomization or patient preference, allowing assessment of outcomes under both controlled and real-world conditions. All procedures are standardized across participating centers, utilizing a two-tunnel fixation technique and augmented with an internal brace (Fibertape) to enhance graft stability.

Outcomes will be assessed over 24 months, including validated patient-reported measures (KOOS, IKDC, Tegner), MRI-based graft evaluation (volume, signal, extrusion, morphology), reoperation rates, complications, satisfaction, and return-to-sport. By integrating randomized comparison with pragmatic elements, this study aims to generate clinically applicable evidence on the relative benefits and limitations of autologous tendon graft versus MAT. The findings are expected to inform surgical decision-making, optimize patient outcomes, and guide future treatment recommendations for young patients suffering from post-meniscectomy syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 45 years

History of partial meniscectomy > 6 months prior to enrollment

Symptomatic post-meniscectomy syndrome (knee pain, swelling, or functional decline)

MRI showing cartilage status ≤ Outerbridge grade 2

Knee joint stability (or stabilized during the index surgery)

Body mass index (BMI) < 30

Willingness to provide written informed consent

Exclusion Criteria:

Tibial slope > 16°

Radiographic or arthroscopic evidence of advanced cartilage degeneration (Outerbridge > 2 or ICRS ≥ 3)

Presence of inflammatory arthritis or systemic inflammatory joint disease

History of cartilage repair surgery

Malalignment > 5° not corrected

Untreated ligamentous instability

Any other condition judged by the investigator to compromise study participation or outcomes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline, 6, 12, and 24 months after surgery (primary analysis at 24 months)
  The KOOS questionnaire evaluates knee-related symptoms, pain, activities of daily living, sports/recreation function, and knee-related quality of life. The primary endpoint is the change in KOOS total score from baseline to 24 months postoperatively.

SECONDARY OUTCOMES:
MRI-Based Graft Evaluation | 12 and 24 months postoperatively
  MRI assessment of graft morphology including volume, signal distribution, shape, and extrusion, evaluated by blinded radiologists
IKDC (International Knee Documentation Committee) Subjective Knee Evaluation | Baseline, 6, 12, and 24 months after surgery
  Patient-reported outcome questionnaire assessing symptoms, daily and sports activities, and knee function
Tegner Activity Scale | Baseline, 6, 12, and 24 months after surgery
  Patient-reported physical activity level, ranging from daily living to competitive sports participation.
Reoperation Rate | Up to 24 months postoperatively
  Incidence of revision surgery or additional procedures related to meniscal reconstruction
Complications | Within 24 months after surgery
  Adverse events related to the surgical intervention, including infection, graft failure, or hardware complications
Patient Satisfaction | 12 and 24 months postoperatively
  Self-reported satisfaction with surgical outcomes, measured using a 5-point Likert scale (very dissatisfied to very satisfied)
Return to Sport Time | Up to 24 months postoperatively
  Time (in months) until patients resume pre-injury level of sports participation, recorded through follow-up interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung memorial hospital, Taoyuan, taoyuan 333, Taoyuan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No
1. Protection of participant privacy and confidentiality is paramount in this study involving sensitive medical data and procedures. Sharing identifiable IPD could breach the trust and privacy of these patients undergoing knee surgeries.
  2. The informed consent process likely did not explicitly state or obtain approval from participants to share their individual-level data, including medical images, functional assessments, and clinical outcomes, with third parties outside the research team.

REFERENCES:
- [Background] Seitz AM, Leiprecht J, Schwer J, Ignatius A, Reichel H, Kappe T. Autologous semitendinosus meniscus graft significantly improves knee joint kinematics and the tibiofemoral contact after complete lateral meniscectomy. Knee Surg Sports Traumatol Arthrosc. 2023 Jul;31(7):2956-2965. doi: 10.1007/s00167-022-07300-z. Epub 2023 Jan 5. PMID 36604322
- [Background] Ronnblad E, Rotzius P, Eriksson K. Autologous semitendinosus tendon graft could function as a meniscal transplant. Knee Surg Sports Traumatol Arthrosc. 2022 May;30(5):1520-1526. doi: 10.1007/s00167-021-06606-8. Epub 2021 Jun 8. PMID 34100999